CLINICAL TRIAL: NCT06849778
Title: A Phase 1, Open-label, Pharmacokinetic Study of TS-172 in Patients on Hemodialysis
Brief Title: An Open-label Pharmacokinetic Study of TS-172 in Patients on Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS172-03-04
Record Dates: First submitted 2025-02-16; First posted 2025-02-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Patients on Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TS-172 (Experimental)
  Interventions: Drug: TS-172

INTERVENTIONS:
Drug: TS-172 — oral administration of TS-172 20 mg

SUMMARY:
A phase 1, open-label, pharmacokinetic study of TS-172 in patients on hemodialysis

ELIGIBILITY:
Inclusion Criteria:

1. Japanese male patients (outpatients) with chronic kidney disease receiving hemodialysis (HD or HDF) 3 times a week for at least 12 weeks prior to the screening test
2. Patients aged >= 18 and < 75 years at the time of obtaining informed consent

Exclusion Criteria:

1. Patients with gastric or intestinal ulceration or a history of them within the past year prior to the date of initiation of treatment, or patients with inflammatory bowel disease or irritable bowel syndrome, or a history of these within the past 5 years prior to the date of initiation of treatment
2. Patients scheduled for renal transplantation, home hemodialysis or change of dialysis facility (transfer or temporary dialysis at other hospital) during the study period
3. Patients who frequently experience diarrhea (defined as Bristol Stool Scale score of 6 or higher)

Ages: 18 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2025-03-22 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Concentration of unchanged form in plasma | Day 1, 2, 8 and 9
Concentration of major metabolites in plasma | Day 1, 2, 8 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No